CLINICAL TRIAL: NCT00309803
Title: Evaluating the Use of the FiberNet® Embolic Protection Device in Carotid Artery Stenting: The EPIC European Study
Brief Title: EPIC European Study: Use of the FiberNet® Emboli Protection Device in Carotid Artery Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumen Biomedical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 872
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid artery; distal protection device
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FiberNet Embolic Protection Device

SUMMARY:
Multicenter, prospective, study designed to demonstrate the performance and safety of the Lumen Biomedical, Inc. FiberNet Embolic Protection System as an adjunctive device during carotid artery percutaneous intervention. The primary endpoint is the rate of all stoke and death within 30 days of the procedure.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to demonstrate the performance and safety of the Lumen Biomedical, Inc. FiberNet® Embolic Protection System as an adjunctive device during carotid artery percutaneous intervention. The feasibility study will involve a maximum of 50 subjects to be enrolled using the FiberNet® during clinically indicated percutaneous intervention of the carotid artery and followed through 30 days post procedure. Subject will be enrolled in up to 5 European Investigational Sites. The study is a prospective multi-center registry with sequential enrollment of qualified subjects who consent to participate and meet all entrance criteria.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for percutaneous stenting with target lesion located within common or internal carotid artery.
* Symptomatic with atherosclerotic stenosis ≥ 50% or asymptomatic with atherosclerotic stenosis ≥ 70% of the carotid artery by NASCET Criteria.
* Targeted vessel diameter for FiberNet placement between 1.75 mm and 7.0 mm.
* The investigator determines that all branch vessels distal to the target lesion and proximal to the proposed site of device deployment will be adequately protected.

Exclusion Criteria:

* Prior stenting of ipsilateral carotid.
* Planned treatment of contralateral carotid within 30 days.
* Experienced a myocardial infarction within the last 14 days.
* Undergone an angioplasty or PTCA/PTA procedure within the past 48 hours.
* Undergone cardiac surgery within the past 60 days.
* Has a planned invasive surgical procedure within 30 days.
* Suffered a stroke within the past 14 days.
* Suffered a transient ischemic neurological attack (TIA) or amaurosis fugax within the past 48 hours.
* Total occlusion of the target vessel.
* Lesions within 2 cm of the ostium of the common carotid artery.
* A stenosis that is known to be unsuitable for stenting because of one or more of: Tortuous or calcified anatomy proximal or distal to the stenosis, Presence of visual thrombus, Pseudo occlusion (string sign).
* Serial lesions that requires more then one stent to cover entire lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
The primary endpoint is the rate of all death and stroke within 30 days of the procedure.

SECONDARY OUTCOMES:
All death, stroke, and myocardial infarction rates; Non-stroke neurological event rates
Technical success rates; Procedural success rates; Access site complication rates

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, Prof. med., Principal Investigator — Andreas-Gruntzig-Haus
Locations (3):
- Germany (3):
  - Dortmund
  - Frankfurt
  - Hamburg